CLINICAL TRIAL: NCT02093325
Title: A Randomized, Double Blind Placebo-controlled Study to Assess the Efficacy and Safety of Eltrombopag as a Rescue of Isolated Chemotherapy-induced Thrombocytopenia in Patients With Solid Tumor
Brief Title: A Study to Assess the Efficacy and Safety of Eltrombopag as a Rescue of Isolated Chemotherapy-induced Thrombocytopenia
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 102-4363A3
Record Dates: First submitted 2014-03-17; First posted 2014-03-21 (Estimated); Last update posted 2017-10-24 (Actual); Status verified 2017-10

CONDITIONS: Solid Tumor
Keywords: eltrombopag , thrombocytopenia, solid tumor
MeSH Terms: conditions — Thrombocytopenia | interventions — eltrombopag

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- eltrombpag (Experimental): Eligible patients will be enrolled randomly in 2:1 ratio to Investigational Drug (Eltrombopag) arm, 50 mg/day, or placebo arm for 7 days.
  Interventions: Drug: Eltrombopag
- Eltrombopag/placebo (Placebo Comparator): Eligible patients will be enrolled randomly in 2:1 ratio to Investigational Drug (Eltrombopag) arm, 50 mg/day, or placebo arm for 7 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Eltrombopag — This will be a Phase III, randomized, double-blind, placebo-controlled clinical trial. Qualified subjects will be randomly assigned to receive either the test treatment or the placebo at 2:1 ratio. Once subjects are randomized, they will be treated with Arm A: Eltrombopag 50 mg/day (n=55) or Arm B: placebo (n=28) once a day for 7 days.
  Other Names: Revolade
  Arms: eltrombpag
Drug: Placebo — This will be a Phase III, randomized, double-blind, placebo-controlled clinical trial. Qualified subjects will be randomly assigned to receive either the test treatment or the placebo at 2:1 ratio. Once subjects are randomized, they will be treated with Arm A: Eltrombopag 50 mg/day (n=55) or Arm B: placebo (n=28) once a day for 7 days.
  Arms: Eltrombopag/placebo

SUMMARY:
The purpose of this study is evaluate the efficacy and safety of eltrombopag as a rescue of isolated chemotherapy-induced thrombocytopenia in patients with solid tumor .

DETAILED DESCRIPTION:
For the phase III study, a double-blind randomized, placebo controlled, parallel-group design will be conducted to evaluate the efficacy of eltombopag . Each subject will be randomly assigned to either Arm A (eltombopag) or Arm B (placebo) in 2:1 ratio.

The primary objective is to compare the response rates of the two treatment arms, Therefore, the two-proportion z test will be considered and sample size can be chosen to achieve an 95% power for detecting a clinically meaningful difference at level of significance=0.05. A difference of 40% in clinical response is considered of clinically meaningful difference between the two treatment arms (75% for eltombopag vs. 35% for placebo). It requires a total sample of 83 subjects (55 for eltombopag and 28 for placebo). According to the 10% loss of screening failure, 90-100 subjects (60-67 for eltombopag and 30-33 for placebo) will be recruited.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged ≥18 years
* Diagnosed with solid tumor
* On active chemotherapy with combined regimen
* A baseline platelet count of <75,000/μL within 2 days of screening
* Hb ≧ 9.0 g/dL
* ANC ≧ 1,500/uL
* GOT and GPT ≤ 3 x ULN
* Serum bilirubin ≤ 1.5 x ULN
* Albumin ≥ 2.5 g/dL
* Adequate renal function for chemotherapy:

serum creatinine ≤ 1.5 × ULN (CTCAE Grade 1).

* Be able to take oral medicine
* ECOG performance ≤ 2
* Has a negative urine or serum pregnancy test at screening and is willing to use contraceptive measures during medication of this trial (Non-childbearing potential is defined as hysterectomy, bilateral oophorectomy, bilateral salpingectomy, tubal ligation and post-menopausal status) for patients with childbearing potential
* Ability to participate and willingness to give written informed consent and to comply with the study restrictions

Exclusion Criteria:

* Single agent chemotherapy or not having chemotherapy
* Serious cardiac, cerebrovascular, or pulmonary disease that, in the opinion of the investigator, would preclude trial medication
* Severe GI tract obstruction that require continuous NG decompression
* Subjects with hemoglobinopathies, e.g. sickle cell anaemia, thalassemia major
* Any prior history of arterial or venous thrombosis
* Any disease condition associated with active bleeding or requiring anticoagulation, heparin or warfarin
* Pre-existing cardiac disease (congestive heart failure New York Heart Association (NYHA) Grade III/IV), (See Appendix 1), or arrhythmias known to involve the risk of thromboembolic events (e.g. atrial fibrillation), or subjects with a QTc >450 msec.
* Seizure disorder that has not been well controlled
* Pregnant or nursing women
* Thyroid dysfunction not adequately controlled.
* Within 2months prior to entering the study, been received radiotherapy to more than 20% bone marrow bearing sites.
* Administration of an investigational drug within 30 days or 5 half-lives, whichever is longer, preceding the first dose of investigational product in the study. Concurrent participation in another interventional clinical trial or administration of any investigational drug during the study is also not permitted.
* A known immediate or delayed hypersensitivity reaction or idiosyncrasy that, in the opinion of the Investigator is due to drugs chemically related to eltrombopag
* Subjects taking anti-neoplastic and immunomodulatory medications (this includes mycophenolate mofetil, thymosine alpha, and extended courses of supraphysiologic doses of steroids)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Estimated)
Dates: Start 2014-03; Primary Completion 2019-03 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
efficacy of eltrombopag (50mg once daily) | up to treatment eltrombopag 7 days
  Evaluate the efficacy of eltrombopag (50mg once daily) compared to the placebo by assessment of response rate

SECONDARY OUTCOMES:
safety and feasibility of 7-day eltrombopag | up to treatment eltrombopag 7 days
  Number of Participants with Chemotherapy-induced thrombocytopenia to assess safety and feasibility to Change from Baseline in use eltrombopag at 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Hung-Hsueh Chou, Principal Investigator — Clinical Trial Center, Chang Gung Memorial Hospital at Linkou
Locations (3):
- Taiwan (3):
  - Department of Obstetrics & Gynecology and Department of Oncology Chang Gung Memorial Hospital, Chiayi City
  - Department of Obstetrics & Gynecology Chang Gung Memorial Hospital, Kaohsiung City
  - Division of Gynecologic Oncology, Department of Obstetrics & Gynecology and Division of Oncology Chang Gung Memorial Hospital, Linkou District